CLINICAL TRIAL: NCT05999864
Title: Efficacy of Proprioceptive Neuromuscular Facilitation Exercise Programme Versus Usual Care in Patients With Total Knee Arthroplasty: A Randomised Controlled Trial
Brief Title: Efficacy of Proprioceptive Neuromuscular Facilitation Exercise Programme in Patients With Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Fatih Ozden, Assistant Professor, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TDAPNF
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Knee Arthroplasty
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): In addition to the program given to the control group, proprioceptive neuromuscular facilitation exercise will be given to the study group as previously described (Gstoettner et al., 2011). These applications will be applied to the patients for 8 weeks, 2 days a week in the clinical environment after the initial evaluation. In addition, both groups will be told that they can contact the researcher when requested.
  Interventions: Other: Rehabilitation
- Control Group (Active Comparator): The control group will receive the usual post-operative care of stretching lower extremity strengthening balance exercises activities of daily living recommendations.
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — Proprioceptive neuromuscular facilitation exercise will be given to the study group as previously described (Gstoettner et al., 2011). These applications will be applied to the patients for 8 weeks, 2 days a week in the clinical environment after the initial evaluation. In addition, both groups will be told that they can contact the researcher when requested.

SUMMARY:
This study was planned to investigate the effectiveness of usual care and proprioceptive neuromuscular facilitation exercise program in patients undergoing total knee arthroplasty surgery. It is aimed to evaluate pain intensity, disability level, proprioception, kinesiophobia, balance, range of motion and functional status of the patients. The study will be conducted with volunteer patients who are followed up by the Orthopedics and Traumatology outpatient clinic of Fethiye State Hospital and who have undergone total knee arthroplasty surgery. The evaluations will be performed in the Orthopedics and Traumatology outpatient clinic of Fethiye State Hospital. It is aimed to evaluate at least 32 patients for the study. The first evaluation will be performed 6 weeks post-operatively and the second evaluation will be performed 2 months after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Having undergone unilateral total knee arthroplasty surgery and being 6 weeks postoperative
* Participate in all necessary follow-up assessments
* 60 years of age or older
* Understand simple commands
* Signing the consent form

Exclusion Criteria:

* A previous history of total knee arthroplasty
* Presence of revision surgery
* Presence of severe osteoarthritis in the contralateral knee
* Severe acute metabolic neuromuscular and cardiovascular diseases
* Extreme obesity (bki>35)
* Presence of malignancy
* Have any other orthopedic or neurological problem that may affect treatment and assessments
* Situations that prevent communication
* Lack of cooperation during the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-06-08 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Change from Baseline VAS at 8 weeks
  On a 10 cm straight line or numeric scale, the patient is asked to mark the pain they feel (0: no pain, 10: excruciating pain).
Western-Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Change from Baseline WOMAC at 8 weeks
  Functionality level in the patient group with knee OA was measured using WOMAC. WOMAC consists of 3 main headings: pain intensity, stiffness and physical function. The individuals included in the study are asked to score each item between 0 (no pain, stiffness, difficulty) and 5 (very severe pain, stiffness, difficulty). The total score ranges from 0 (no disability) to 96 (complete disability).
Knee Joint Proprioception Measurement | Change from Baseline Knee Joint Proprioception Measurement at 8 weeks
  The inclinometer is placed distal to the tibial tuberosity. In full knee extension, the patient is asked to perform a single leg squat with eyes closed or unable to see the leg being tested. He/she is allowed to support with his/her hands to prevent loss of balance. When the knee flexion angle of 30° is reached, the patient is asked to stop and stay at this point for 5 seconds. Then return to full knee extension. This movement is repeated 3 times. This time, without any stop command, the patient is asked to reach the same 30° knee flexion angle as in the previous exercises. This application is also repeated 3 times. The "absolute angle difference", which is the difference between the targeted angle in each repetition and the angle realized by the patient, is recorded. The arithmetic mean of the 3 repetitions' absolute angle difference is recorded as the result data.
Modified Four Square Step Test (mFSST) | Change from Baseline mFSST at 8 weeks
  A suitable background is divided into four identical squares with a "+" shaped line using tape. The squares are numbered with numbers between 1-4 in a clockwise direction and this sequence is explained to the participant. The patient steps from the starting point to squares 1,2,3 and 4 in a way that the direction remains the same and without stepping on the lines. The test is terminated when the last foot contact is interrupted at square 4. The time elapsed during the main measurement is recorded with a stopwatch.
Figure 8 Walking Test (F8WT) | Change from Baseline F8WT at 8 weeks
  Participants are instructed to stand at the midpoint between two cones (1.52 m apart) and look at one of the cones. Participants are asked to walk in a circle of 8 around the cones at a comfortable speed and direction of their choice. The stopwatch is stopped while returning to the starting point. The elapsed time and the number of steps taken are recorded.
Berg Balance Scale (BBS) | Change from Baseline BBS at 8 weeks
  The 14 items in the scale assess static sitting and standing balance as well as expected balance during activities. Scoring is done on a 5-point scale that takes into account whether the patient can perform the task safely and independently and is usually based on a specific time interval. Normal performances are rated from 0 (unable to perform) to 4 points (normal performance). Scores on individual items are summed for a total score, with a maximum score of 56 points.
Activity Specific Balance Confidence Scale (ABC) | Change from Baseline ABC at 8 weeks
  This scale includes 16 tasks related to indoor and outdoor activities of daily living to measure balance confidence in older people with various levels of function. Scores for each question range from 0% (no confidence) to 100% (full confidence). Higher scores indicate greater confidence.
Tampa Scale for Kinesiophobia (TSK) | Change from Baseline TSK at 8 weeks
  The questionnaire is a 17-item scale developed to measure fear of movement/reinjury. The normal score range is between 17 and 68.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Özden, PhD, Study Director — Muğla Sıtkı Koçman University
Locations (1):
- Muğla, Muğla, Turkey (Türkiye)